CLINICAL TRIAL: NCT00009854
Title: Phase I/II Study of Intratumoral Injection of DTI-015 Prior to Tumor Resection in Patients With Recurrent Malignant Glioma or Metastatic Neoplasm to Brain
Brief Title: Carmustine Followed By Surgery in Treating Patients With Recurrent Supratentorial Malignant Glioma or Metastatic Brain Neoplasm
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Direct Therapeutics (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068416; DTI-0002; UCSF-H7858-17520-01; NCI-V00-1642
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2003-03

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer
Keywords: adult glioblastoma; tumors metastatic to brain; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Glioblastoma; Brain Neoplasms; Astrocytoma; Ependymoma; Oligodendroglioma; Gliosarcoma | interventions — Carmustine; Ethanol

INTERVENTIONS:
Drug: carmustine in ethanol
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of carmustine followed by surgery in treating patients who have recurrent supratentorial malignant glioma or metastatic brain neoplasm.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the extent and pattern of distribution of DNA adducts in patients with recurrent supratentorial malignant glioma or metastatic neoplasm to the brain treated with neoadjuvant intratumoral carmustine in ethanol (DTI-015) followed by tumor resection.
* Determine the qualitative and quantitative toxicity of this treatment regimen in these patients.

OUTLINE: This is a dose escalation study.

Patients receive neoadjuvant carmustine in ethanol (DTI-015) intratumorally under stereotactic guidance 45-90 minutes prior to craniotomy and tumor resection.

Cohorts of 3-6 patients receive escalating doses of DTI-015 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 3 or 3 of 6 patients experience dose-limiting toxicity.

Patients are followed at 4, 8, and 12 weeks, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent supratentorial malignant glioma with clear evidence of progression by MRI

  * Glioblastoma multiforme
  * Anaplastic ependymoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma OR
* Metastatic tumor to the brain other than melanoma
* Planned resection of tumor (must be first surgery for recurrent disease)
* Tumor volume of each tumor component or residual tumor must be at least 4 cm3 and no greater than 33.4 cm3
* Tumor shape and surrounding structure(s) unlikely to cause an irregular distribution of the injected study drug

  * Tumor is spherical, spheroid, or ovoid
  * No tumors shaped into 3 or more components (e.g., multicentric or multilobulated)
  * No tumors extending into the ventricular system
  * Tumor has an intact stroma (i.e., tumor mass not partially incised or punctured)
  * Central necrosis and/or central cystic areas allowed if an enhancing rim with a thickness of more than 5 mm is present
* No tumors in the following locations of the brain:

  * Brainstem (pons or medulla)
  * Midbrain (mesencephalon)
  * Primary sensorimotor cortex in the dominant hemisphere
  * Within 1.5 cm of the optic chiasm, either optic nerve, or any other cranial nerve

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No evidence of bleeding diathesis

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT and SGPT no greater than 2.5 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 40 mL/min OR
* BUN no greater than 30 mg/dL

Other:

* No active uncontrolled infection
* Afebrile (37.5 degrees C) unless fever due to tumor
* No other unstable or severe medical condition
* No complicating medical or psychiatric problem that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior systemic chemotherapy (6 weeks for nitrosoureas, mitomycin, or Gliadel wafers) and recovered
* No anti-tumor chemotherapy within 12 weeks after study drug unless tumor volume increases by more than 25% by MRI

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No prior intracranial brachytherapy
* No anti-tumor radiotherapy within 12 weeks after study drug unless tumor volume increases by more than 25% by MRI

Surgery:

* See Disease Characteristics
* Prior surgery allowed
* No anti-tumor surgery within 12 weeks after study drug

Other:

* No concurrent anticoagulants
* No other concurrent investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Gene David Resnick, MD, Study Chair — Millennix
Locations (2):
- United States (2):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Massey Cancer Center, Richmond, Virginia